CLINICAL TRIAL: NCT02840396
Title: Role of Executive Function in Language: an Experimental and Clinical Approach With Application to Mother Language and Second Language
Brief Title: Effect of rTMS of the Dorsolateral Prefrontal Cortex on Language Production in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Marie Annoni (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor-Investigator, Jean-Marie Annoni, Prof. Dr. med., University of Fribourg
Organization: University of Fribourg (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SNF325130_156937_2
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Language
Keywords: language; DLPFC; rTMS; Executive Functions
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS (Experimental)
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator)
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — repetitive TMS (rTMS) can lead to temporary increases or decreases (depending on the protocol used) in excitability of the targeted area. This change in excitability has been shown to last beyond the duration of the stimulation.
  Arms: rTMS
Device: Sham rTMS — Sham rTMS (or placebo rTMS) refers to a control condition in which no physiological effect on the targeted cortical region occurs.
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to investigate the effects of repetitive transcranial magnetic stimulation (rTMS) over the dorsolateral prefrontal cortex (DLPFC) on language production.

DETAILED DESCRIPTION:
Background:

Several studies investigating healthy or clinical populations have shown that (r)TMS applied over the dorsolateral prefrontal cortex (DLPFC) has an effect on language-related processes such as verbal working memory (Osaka et al., 2007), sentence comprehension (Cotelli et al., 2011) and language switching (Holtzheimer et al., 2005, Nardone et al., 2011).

Clinical observations and neuroimaging studies seem to confirm the role of executive functions and frontal structures in language processing in monolingual and bilingual subjects (e.g. Fabbro et al., 2000, Abutalebi & Green 2007). However, only few studies investigated the effects of modulation of cognitive control-networks on lexical access.

Aim and procedure:

The study will investigate the role of the DLPFC and executive functioning in L1 and L2 language processing. The core question is whether rTMS over the DLPFC will influence lexical access and language production.

Each participant will take part in two sessions: 1. rTMS session 2. Sham rTMS session. After the application of rTMS/Sham rTMS, the participants will conduct two language tasks (translation, picture naming) and a non-verbal task, while the EEG is recorded.

ELIGIBILITY:
Inclusion Criteria:

* L1 French, knowledge of English as a foreign language
* 18-45 years of age
* Right-handedness

Exclusion Criteria:

* epilepsy /family history of epilepsy
* brain surgery, traumatic brain injuries
* cardiac pacemaker, metallic objects in the body
* history of neurological diseases or psychiatric disorders
* drug use (alcohol, psychoactive medication)
* developmental language disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Language production | within 30 mins after rTMS/sham rTMS
  Picture naming task and word translation task

SECONDARY OUTCOMES:
non-verbal executive functions task | within 30 mins after rTMS/sham rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Annoni, Prof. Dr., Principal Investigator — University of Fribourg
Locations (1):
- Laboratory for Cognitive and Neurological Sciences, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osaka N, Otsuka Y, Hirose N, Ikeda T, Mima T, Fukuyama H, Osaka M. Transcranial magnetic stimulation (TMS) applied to left dorsolateral prefrontal cortex disrupts verbal working memory performance in humans. Neurosci Lett. 2007 May 18;418(3):232-5. doi: 10.1016/j.neulet.2007.01.087. Epub 2007 Apr 8. PMID 17467169
- [Background] Cotelli M, Calabria M, Manenti R, Rosini S, Zanetti O, Cappa SF, Miniussi C. Improved language performance in Alzheimer disease following brain stimulation. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):794-7. doi: 10.1136/jnnp.2009.197848. Epub 2010 Jun 23. PMID 20574108
- [Background] Holtzheimer P, Fawaz W, Wilson C, Avery D. Repetitive transcranial magnetic stimulation may induce language switching in bilingual patients. Brain Lang. 2005 Sep;94(3):274-7. doi: 10.1016/j.bandl.2005.01.003. PMID 16098377
- [Background] Nardone R, De Blasi P, Bergmann J, Caleri F, Tezzon F, Ladurner G, Golaszewski S, Trinka E. Theta burst stimulation of dorsolateral prefrontal cortex modulates pathological language switching: A case report. Neurosci Lett. 2011 Jan 10;487(3):378-82. doi: 10.1016/j.neulet.2010.10.060. Epub 2010 Oct 29. PMID 21036201
- [Background] Fabbro F, Skrap M, Aglioti S. Pathological switching between languages after frontal lesions in a bilingual patient. J Neurol Neurosurg Psychiatry. 2000 May;68(5):650-2. doi: 10.1136/jnnp.68.5.650. PMID 10766900
- [Background] Abutalebi J, Green D. Bilingual language production: The neurocognition of language representation and control. Journal of Neurolinguistics, 20, 242-275, 2007.